CLINICAL TRIAL: NCT05050331
Title: Effectiveness of Muscle Energy Technique and Trigger Point Release in Plantar Fasciitis: a Comparative Study
Brief Title: Comparative Effectiveness of Muscle Energy Technique and Trigger Point Release in Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Faisalabad (Other)
Responsible Party: Principal Investigator, Dr Izza Ayub; PT, Principal Investigator, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TUF/DR/MSPP/174
Record Dates: First submitted 2021-09-02; First posted 2021-09-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Plantar Fasciitis
Keywords: Muscle Energy Technique; Trigger Point Release
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Muscle Energy Technique (MET) Group (Experimental): The MET protocol consisted of post-isometric relaxation applied to the gastrocnemius and soleus muscles, with 5 repetitions per set, 3 times a week, for 4 weeks
  Interventions: Procedure: Muscle Energy Technique; Procedure: Self-Stretching of Calf and Plantar Fascia
- Trigger Point Release Group (Experimental): The gastrocnemius muscle was subjected to trigger point release therapy, 3 sessions per week, over a period of 4 weeks
  Interventions: Procedure: Trigger Point Release; Procedure: Self-Stretching of Calf and Plantar Fascia

INTERVENTIONS:
Procedure: Muscle Energy Technique — MET involves patient-generated muscle contractions 10-20% maximum voluntary contraction from a specific position and direction, resisted by the therapist to facilitate muscle relaxation and lengthening
  Arms: Muscle Energy Technique (MET) Group
Procedure: Trigger Point Release — Trigger point release involved applying 90 seconds of sustained thumb pressure to the trigger point, repeated three times with 30-second relaxation intervals, followed by three caudal-to-cranial longitudinal strokes along the taut band.
  Arms: Trigger Point Release Group
Procedure: Self-Stretching of Calf and Plantar Fascia — Participants performed a self-stretching program, comprising 5 repetitions of 20 seconds of stretching and 20 seconds of relaxation, twice daily

SUMMARY:
This study aimed to investigate the comparative efficacy of Muscle Energy Technique (MET) and Trigger Point Release in the treatment of Plantar Fasciitis. A single-blinded, randomized clinical trial was conducted, wherein thirty participants were randomly assigned to two parallel groups. One group received MET, while the other received Trigger Point Release, with both groups performed self-stretching exercises as part of their home program. Outcome measures included pain intensity and foot function. Treatments were administered three times a week for a duration of four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral plantar heel pain that worsens with weight-bearing activities
* Age range: 25-45 years
* Pain exacerbation with initial morning ambulation (i.e., walking a few steps)
* Presence of at least one identifiable trigger point in the calf muscles

Exclusion Criteria:

* Bilateral heel pain
* History of tumors in the leg or foot
* Previous lower limb fractures
* Recent or unresolved lower limb injuries
* Achilles Tendinitis
* Ankle arthritis
* Surgery
* Vascular Disease

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Foot Pain | Four Weeks
  Numeric Pain Rating Scale served as the primary outcome measure, with decreasing values indicating improved patient condition and reduced pain intensity

SECONDARY OUTCOMES:
Foot Function | Four Weeks
  Foot function index was utilized as a secondary outcome measure, with decreasing scores indicating improved foot function and reduced functional impairment as patient condition improves

CONTACTS AND LOCATIONS:
Overall Officials: Dr Sidra Majeed; PT, MSPP, Study Director — The University of Faisalabad
Locations (1):
- The University of Faisalabad, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No